CLINICAL TRIAL: NCT01855165
Title: The Role of Clinical Pharmacist's Intervention in Management of Clinically Relevant Drug-drug Interactions in Patients With Chronic Heart Failure
Brief Title: The Role of Clinical Pharmacist in Management of DDIs in CHF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CHF42013; 109/01/13 (Other: National Medical Ethics Committee of the Republic of Slovenia (NMEC))
Record Dates: First submitted 2013-05-06; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; drug-drug interactions; pharmacist's intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advice on DDIs (Experimental): Attending physician will be randomly assigned to intervention arm care as usual; in the intervention arm, he/she will receive advice about DDIs between medications prescribed to patients on top of general heart failure advice.
  Interventions: Behavioral: Advice on DDIs
- General advice (No Intervention)

INTERVENTIONS:
Behavioral: Advice on DDIs
  Arms: Advice on DDIs

SUMMARY:
Drug-drug interactions (DDIs) are common in patients with chronic heart failure (CHF) and their incidence increases with the number of drugs that the patients are prescribed for treatment of their condition. Data bases often detect DDIs that are of high clinical relevance. The investigators have performed this study in order to detect clinically significant DDIs and to diminish their occurrence by sending notification about DDIs to attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with diagnosis of CHF I50.0 - I50.9 and I11.0 - I11.9 (ICD-10)
* patients treated with at least two drugs

Exclusion Criteria:

* Patients admitted to other conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To assess the difference in frequency and severity of clinically significant DDIs in control arm and interventional arm between admission and discharge | 90 days
  We will measure the difference in clinically significant DDIs between admission and discharge. The doctors in control group will not receive the advice about DDIs between drugs prescribed to patient, while the doctors in interventional group will. With this will will assess the impact of the advice in the occurence of DDIs between admission and discharge for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainscak, PhD, Principal Investigator — University Clinic Golnik
Locations (1):
- University Clinic Golnik, Golnik, Slovenia

REFERENCES:
- [Derived] Roblek T, Deticek A, Leskovar B, Suskovic S, Horvat M, Belic A, Mrhar A, Lainscak M. Clinical-pharmacist intervention reduces clinically relevant drug-drug interactions in patients with heart failure: A randomized, double-blind, controlled trial. Int J Cardiol. 2016 Jan 15;203:647-52. doi: 10.1016/j.ijcard.2015.10.206. Epub 2015 Oct 28. PMID 26580349